CLINICAL TRIAL: NCT02127775
Title: A Phase 1, Randomized, Open-Label, Crossover Study to Assess the Bioequivalence of Lesinurad Tablets From Two Manufacturing Sites in Healthy Adult Male Subjects
Brief Title: Lesinurad Tablet Bioequivalence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-132
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence B (Experimental): Day 1: Lesinurad 400 mg (manufactured at Site 2); Day 5: Lesinurad 400 mg (manufactured at Site 1)
  Interventions: Drug: Lesinurad 400 mg (manufactured at Site 1); Drug: Lesinurad 400 mg (manufactured at Site 2)
- Sequence A (Experimental): Day 1: Lesinurad 400 mg (manufactured at Site 1); Day 5: Lesinurad 400 mg (manufactured at Site 2)
  Interventions: Drug: Lesinurad 400 mg (manufactured at Site 1); Drug: Lesinurad 400 mg (manufactured at Site 2)

INTERVENTIONS:
Drug: Lesinurad 400 mg (manufactured at Site 1)
Drug: Lesinurad 400 mg (manufactured at Site 2)

SUMMARY:
This study will assess the bioequivalence of lesinurad tablets manufactured at two different sites.

DETAILED DESCRIPTION:
This study is intended to evaluate the clinical comparability of lesinurad tablets manufactured at the 2 different sites by assessing relevant clinical Pharmacokinetics (PK) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 40 kg/m2.
* Subject has a Screening serum urate level ≤ 7 mg/dL. ˗ Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Subject has any gastrointestinal disorder that affects motility and/or absorption.
* Subject has a history or suspicion of kidney stones.
* Subject has undergone major surgery within 3 months prior to Screening.
* Subject has donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to the Screening visit.
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
PK profile of lesinurad from plasma | Day 1 and Day 5
  PK endpoints in terms of maximum observed concentration (Cmax); time of occurrence of maximum observed concentration (tmax); area under the plasma concentration time curve from zero to 24 hours post dose (AUC last) and from zero to infinity (AUC ∞); and apparent terminal half-life (t1/2). Point estimates and 90% confidence intervals for the ratio of geometric means for Cmax, AUC last and AUC∞ between test and reference formulations.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 5 weeks
  Changes in Laboratory, Electrocardiogram and Vital Signs Parameters

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Austin, Texas, United States